CLINICAL TRIAL: NCT00791570
Title: Histocompatibility Leukocyte Antigen (HLA)-A*2402 and A*0201 Restricted Peptide Vaccine Therapy in Patients With Neovascular Maculopathy
Brief Title: Anti-VEGFR Vaccine Therapy in Treating Patients With Neovascular Maculopathy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Osaka University (Other)
Collaborators: Human Genome Center, Institute of Medical Science, University of Tokyo (Other)
Responsible Party: Yasuo Tano, Department of Ophthalmology, Osaka University Medical School
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08062
Record Dates: First submitted 2008-10-31; First posted 2008-11-14 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Neovascular Maculopathy; Age Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Receptor Protein-Tyrosine Kinases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental)
  Interventions: Biological: VEGFR1 and VEGFR2

INTERVENTIONS:
Biological: VEGFR1 and VEGFR2 — Biological: VEGFR1 and VEGFR2 Patients will be vaccinated once a week for 12 weeks. On each vaccination day, VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection.
  Other Names: VEGFR1; VEGFR2; AMD

SUMMARY:
The purpose of this study is to evaluate the safety and time to progression of HLA-A*2402 or A*0201 restricted epitope peptides VEGFR1 and VEGFR2 emulsified with Montanide ISA 51 in patients with Neovascular Maculopathy, including Age Related Macular Degeneration

DETAILED DESCRIPTION:
VEGF receptor 1 and 2 are essential targets to pathogenic angiogenesis, and we identified that peptides derived from these receptors significantly induce the effective tumor specific CTL response in vitro and vivo. According to these findings, in this trial, we evaluate the safety, immunological and clinical response of those peptides. Patients will be vaccinated once a week for 12 weeks. On each vaccination day, VEGFR1 peptide (1mg) and VEGFR2 peptide (1mg) mixed with Montanide ISA 51 will be administered by subcutaneous injection. In the study, our primary aim is to evaluate the safety and tolerability of these peptide vaccine. The second aim is evaluate the immunological and clinical response of this vaccine therapy.

ELIGIBILITY:
Inclusion Criteria:

* Neovascular Maculopathy including Age Related Macular Degeneration.
* Resistant against PDT or Anti VEGF therapy or Patient disagree with these therapies.
* with HLA-A*2402 or A*0201

Exclusion Criteria:

* Pregnancy(woman of childbearing potential:Refusal or inability to use effective means of contraception) Breastfeeding Active or uncontrolled infection Unhealed external wound Concurrent treatment with steroids or immunosuppressing agent Uncontrolled brain and/or intraspinal lesion(s) Decision of unsuitableness by principal investigator or physician-in-charge

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-10; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Safety of this trial will be assessed based on National Cancer Institute-Common Toxicity Criteria,(NCI-CTC) version3. In case grade 4 or more complications occur, we will report the case to the review board within 14 days. | 3 months

SECONDARY OUTCOMES:
Efficacy of the trail will be assessed by external judge board using fluorescent and ICG angiography and optical coherence tomography. The best corrected visual acuity will be measured before and 3 month after the trail. | 3 month
To evaluate immunological responses. INF-r production of monocytes from the patients after the peptide stimulation will be measured by ELISA. | 3 month

CONTACTS AND LOCATIONS:
Overall Officials: Kohji Nishida, MD, PhD, Study Chair — Chair of Ophthalmology, Osaka University Medical School
Locations (1):
- Ophthalmology, Osaka University Medical School, Suita, Osaka, Japan